CLINICAL TRIAL: NCT04159870
Title: Rifaximin Versus Norfloxacin in the Primary Prophylaxis of Spontaneous Bacterial Peritonitis
Brief Title: Rifaximin Versus Norfloxacin in Spontaneous Bacterial Peritonitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ospedali Riuniti di Foggia (Other)
Responsible Party: Principal Investigator, Antonio Facciorusso, Principal Investigator, Ospedali Riuniti di Foggia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RIFA01
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Rifaximin; Norfloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Rifaximin 1200 mg/day in 3 doses
  Interventions: Drug: Rifaximin
- Control Group (Active Comparator): Norfloxacin 400 mg/day in one dose
  Interventions: Drug: Norfloxacin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin pills 400 mg x 3/day
  Arms: Intervention Group
Drug: Norfloxacin — Norlfloxacin 400 mg 1 pill/day
  Arms: Control Group

SUMMARY:
Background

Prophylaxis of SBP is indicated in three high-risk populations: patients with acute gastrointestinal hemorrhage, patients with low total protein content in ascitic fluid, and patients with a previous history of SBP (secondary prophylaxis).

Selective intestinal decontamination with norfloxacin, a quinolone with relatively poor gastrointestinal absorption and with antibacterial activity against GNB, is the most commonly used regimen, but several concerns have been recently raised in this regard.

A recent network meta-analysis published by the investigators showed that rifaximin determines interesting results in this setting but needs to be tested in further trials.

Given its favorable safety profile and the relatively low cost, rifaximin could represent the antibiotic of choice in long-term prophylaxis.

Study Objective To establish the prophylactic efficacy, of rifaximin as compared to norfloxacin in cirrhotic patients with low protein content in the ascitic fluid.

Protocol design Phase III, two-arms, open-label, multi-center, randomized controlled trial.

Trial population Patients with cirrhosis and ascites and with low protein content in the ascitic fluid (≤1.5 g/dL) and with deteriorated liver function (Child-Pugh score ≥B9, serum bilirubin level ≥3 mg/dL) or impaired renal function (creatinine ≥1.2 mg/dL blood urea nitrogen level ≥25 mg/dL or hyponatremia ≤130 milliequivalent [mEq]/L)

Protocol Treatments

* The Treatment arm will undergo rifaximin 1200 mg/day in 3 doses.
* The Control arm will undergo norfloxacin 400 mg 1/die for 6 months

Primary Endpoint Prevention of spontaneous bacterial peritonitis episodes.

Secondary Endpoints

* Prevention of mortality (both all-cause and liver-related mortality)
* Preventions of hepatorenal syndrome
* Prevention of other infections
* Adverse events

Sample size and study duration It will be planned to enroll 322 patients (161 per arms) within 18 months. A minimum follow up of 6 months from the last patient recruited will be required.

DETAILED DESCRIPTION:
Background

Spontaneous bacterial peritonitis (SBP) is a commonly observed and severe complication in patients with cirrhosis and ascites, with a reported prevalence ranging from 10% to 25% in hospitalized cirrhotic patients1.

Given the high mortality rate and the risk of developing hepato-renal syndrome (HRS), prophylaxis of SBP is indicated particularly in three high-risk populations: patients with acute gastrointestinal hemorrhage, patients with low total protein content in ascitic fluid, and patients with a previous history of SBP (secondary prophylaxis)2.

The ideal prophylactic agent should be safe, affordable, and effective particularly against anaerobic bacteria translocating from the gut as most episodes of SBP are thought to result from the translocation of enteric Gram-negative bacilli (GNB)3.

Selective intestinal decontamination with norfloxacin, a quinolone with relatively poor gastrointestinal absorption and with antibacterial activity against GNB, is the most commonly used regimen4, but several concerns have been recently raised in this regard. In fact, the epidemiology of bacterial infections in cirrhosis is evolving with an increasing incidence of infections caused by quinolone-resistant bacteria5; moreover, primary prophylaxis in low-protein ascitic patients requires long-term antibiotic regimens (whose exact duration is still matter of debate), hence less expensive and better tolerated agents such as rifaximin have been tested with conflicting results6.

A recent network meta-analysis published by the investigators showed that rifaximin determines interesting results in this setting but needs to be tested in further trials7.

Given its favorable safety profile and the relatively low cost, rifaximin could represent the antibiotic of choice in long-term prophylaxis.

Study Objective To establish the prophylactic efficacy, of rifaximin as compared to norfloxacin in cirrhotic patients with low protein content in the ascitic fluid.

Protocol design Phase III, two-arms, open-label, multi-center, randomized controlled trial.

Trial population Patients with cirrhosis and ascites and with low protein content in the ascitic fluid (≤1.5 g/dL) and with deteriorated liver function (Child-Pugh score ≥B9, serum bilirubin level ≥3 mg/dL) or impaired renal function (creatinine ≥1.2 mg/dL blood urea nitrogen level ≥25 mg/dL or hyponatremia ≤130 mEq/L)

Protocol Treatments

* The Treatment arm will undergo rifaximin 1200 mg/day in 3 doses.
* The Control arm will undergo norfloxacin 400 mg 1/die for 6 months

Protocol

Baseline evaluation will include history and physical examination, liver and renal tests, ascitic fluid analysis and culture, fresh urine sediment, and abdominal ultrasonography. Treatment will start immediately after randomization. Follow-up visits will be performed every 4 weeks. Treatment compliance will be assessed by interviewing the patient and by tablet count at each visit. A patient will be considered noncompliant when the study medication will not be taken for 7 days or more, or will fail to take more than 20 % of their pills or miss two or more visits.

Medications will be interrupted when patients develop an episode of SBP (ascitic fluid neutrophil count[ 250 cell/ml with or without clinical evidence), or have upper gastrointestinal (GIT) bleeding or receive a liver transplant.

Diagnostic paracentesis will be performed when clinically indicated. Diagnosis of spontaneous bacteremia, SBP, urinary infection, and other infections will be made by biological fluid cultures and analysis; type-1 and type-2 HRS will be diagnosed according to the criteria of the International Ascites Club. Spontaneous bacteremia and SBP will be treated with ceftriaxone.

Primary Endpoint Prevention of spontaneous bacterial peritonitis episodes.

Secondary Endpoints

* Prevention of mortality (both all-cause and liver-related mortality)
* Preventions of hepatorenal syndrome
* Prevention of other infections
* Adverse events

Sample size and study duration It will be planned to enroll 322 patients (161 per arms) within 18 months. A minimum follow up of 6 months from the last patient recruited will be required.

Treatment strategy Patients complying with the eligibility criteria will be randomized in a 1:1 fashion to receive rifaximin 1200 mg/day or norfloxacin 400 mg/day. No cross-over will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with cirrhosis and ascites and with low protein content in the ascitic fluid (≤1.5 g/dL) and with deteriorated liver function (Child-Pugh score ≥B9, serum bilirubin level ≥3 mg/dL) or impaired renal function (creatinine ≥1.2 mg/dL blood urea nitrogen level ≥25 mg/dL or hyponatremia ≤130 mEq/L)

Exclusion Criteria:

* Age under 18 years
* Previous history of SBP
* Previous use of antibiotics within the previous two weeks
* Previous GIT bleeding within one month
* Resolving ascites for one month after diuretic therapy
* Liver malignancy, organic renal disease
* Human immunodeficiency virus infection
* Known hypersensitivity to planned drugs
* Refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Prevention of Spontaneous Bacterial Peritonitis | 6 months
  Rate of episodes of spontaneous bacterial peritonitis

SECONDARY OUTCOMES:
Prevention of mortality | 6 months
  Rate of deaths observed
Prevention of hepatorenal syndrome | 6 months
  Rate of hepatorenal syndrome episodes
Prevention of other infections | 6 months
  Rate of other infections
Adverse Events | 6 months
  Rate of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedali Riuniti Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fernandez J, Navasa M, Gomez J, Colmenero J, Vila J, Arroyo V, Rodes J. Bacterial infections in cirrhosis: epidemiological changes with invasive procedures and norfloxacin prophylaxis. Hepatology. 2002 Jan;35(1):140-8. doi: 10.1053/jhep.2002.30082. PMID 11786970
- [Result] European Association for the Study of the Liver. EASL clinical practice guidelines on the management of ascites, spontaneous bacterial peritonitis, and hepatorenal syndrome in cirrhosis. J Hepatol. 2010 Sep;53(3):397-417. doi: 10.1016/j.jhep.2010.05.004. Epub 2010 Jun 1. No abstract available. PMID 20633946
- [Result] Piano S, Brocca A, Mareso S, Angeli P. Infections complicating cirrhosis. Liver Int. 2018 Feb;38 Suppl 1:126-133. doi: 10.1111/liv.13645. PMID 29427501
- [Result] Soriano G, Guarner C, Tomas A, Villanueva C, Torras X, Gonzalez D, Sainz S, Anguera A, Cusso X, Balanzo J, et al. Norfloxacin prevents bacterial infection in cirrhotics with gastrointestinal hemorrhage. Gastroenterology. 1992 Oct;103(4):1267-72. doi: 10.1016/0016-5085(92)91514-5. PMID 1397884
- [Result] Aparicio JR, Such J, Pascual S, Arroyo A, Plazas J, Girona E, Gutierrez A, de Vera F, Palazon JM, Carnicer F, Perez-Mateo M. Development of quinolone-resistant strains of Escherichia coli in stools of patients with cirrhosis undergoing norfloxacin prophylaxis: clinical consequences. J Hepatol. 1999 Aug;31(2):277-83. doi: 10.1016/s0168-8278(99)80225-6. PMID 10453941
- [Result] Menshawy A, Mattar O, Barssoum K, AboEl-Naga AM, Salim HM, Mohamed AMF, Elgebaly A, Abd-Elsalam S. Safety and Efficacy of Rifaximin in Prophylaxis of Spontaneous Bacterial Peritonitis: A Systematic Review and Meta-analysis. Curr Drug Targets. 2019;20(4):380-387. doi: 10.2174/1389450119666180924145156. PMID 30246636
- [Result] Facciorusso A, Papagiouvanni I, Cela M, Buccino VR, Sacco R. Comparative efficacy of long-term antibiotic treatments in the primary prophylaxis of spontaneous bacterial peritonitis. Liver Int. 2019 Aug;39(8):1448-1458. doi: 10.1111/liv.14109. Epub 2019 Apr 25. PMID 30920712
- [Result] Goel A, Rahim U, Nguyen LH, Stave C, Nguyen MH. Systematic review with meta-analysis: rifaximin for the prophylaxis of spontaneous bacterial peritonitis. Aliment Pharmacol Ther. 2017 Dec;46(11-12):1029-1036. doi: 10.1111/apt.14361. Epub 2017 Oct 9. PMID 28994123
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180